| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | ÷ | Open-Label, Single-Sequence Study to Evaluate the Effects of Darunavir/Ritonavir and/or Etravirine on the Pharmacokinetics of GSK3640254 and the Effects of GSK3640254 on the Pharmacokinetics of Darunavir/Ritonavir and/or Etravirine in Heathy Adults |
| <b>Compound Number</b> | : | GSK3640254 |
| <b>Effective Date</b> | : | 15/10/2021 |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report (CSR) for Protocol 213054.
- This RAP is intended to describe the full analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRODUC | CTION | 4 |
| 2. | <ul><li>2.1. Cha</li><li>2.2. Stud</li><li>2.3. Stud</li><li>2.4. Stat</li></ul> | OF KEY PROTOCOL INFORMATION anges to the Protocol Defined Statistical Analysis Plan dy Objective(s) and Endpoint(s). dy Design tistical Hypotheses mple Size Determination | 4<br>6<br>7 |
| 3. | | ANALYSESal Analyses | |
| 4. | | POPULATIONStocol Deviations | |
| 5. | CONVENT<br>5.1. Stud<br>5.2. Bas<br>5.3. Oth | RATIONS FOR DATA ANALYSES AND DATA HANDLING TIONS | 10<br>10 |
| 6. | | PPULATION ANALYSESerview of Planned Study Population Analyses | |
| 7. | 7.1. Prin | 3. Population of Interest | |
| | 7.2. Sec<br>7.2.<br>7.2.<br>7.2.<br>7.2.<br>7.2. | condary Pharmacokinetic Analyses 1. Endpoint / Variables 1. 7.2.1.1. Drug Concentration Measures 1. Summary Measure 1. Population of Interest | 15<br>15<br>15<br>15 |
| 8. | 8.1. Adv<br>8.2. Clin<br>8.3. Adv<br>8.4. Oth | NALYSES verse Events Analyses nical Laboratory Analyses verse Events of Special Interest er Safety Analyses VID 19 Related Analyses | 17<br>17<br>17 |
| 9 | REFERENC | CES | 19 |


| 213054 |
|----------|
| 713115/1 |

| 10. | <b>APPE</b> | NDICES | | 20 |
|---|---|---|---|---|
| | 10.1. | Appendi | x 1: Schedule of Activities | 20 |
| | | 10.1.1. | Protocol Defined Schedule of Events | 20 |
| | 10.2. | Appendi | x 2: Study Phases and Treatment Emergent Adverse | |
| | | Events | | 35 |
| | | 10.2.1. | | 35 |
| | | | 10.2.1.1. Study Phases for Lab, Electrocardiograms, and | |
| | | | Vital Signs | |
| | | | 10.2.1.2. Study Phases for Concomitant Medication | |
| | | 10.2.2. | Treatment Emergent Flag for Adverse Events | |
| | 10.3. | | x 3: Data Display Standards & Handling Conventions | |
| | | 10.3.1. | Reporting Process | |
| | | 10.3.2. | Reporting Standards | |
| | | 10.3.3. | Reporting Standards for Pharmacokinetics | |
| | 10.4. | | x 4: Derived and Transformed Data | |
| | | 10.4.1. | General | |
| | | 10.4.2. | Study Population | |
| | | 10.4.3. | Safety | |
| | 10.5. | | x 5: Reporting Standards for Missing Data | |
| | | | Premature Withdrawals | |
| | | 10.5.2. | | |
| | | | 10.5.2.1. Handling of Missing and Partial Dates | 41 |
| | 10.6. | Appendi | x 6: Division of AIDS (DAIDS) Table for Grading the | |
| | | | of Adult and Pediatric Adverse Events | |
| | | | Laboratory Values | |
| | 10.7. | | x 7: Values of Potential Clinical Importance | |
| | | | ECG | |
| | | | Vital Signs | |
| | 10.8. | | x 8: Abbreviations & Trademarks | |
| | | 10.8.1. | | |
| | 40.0 | 10.8.2. | | |
| | 10.9. | | x 9: List of Data Displays | |
| | | 10.9.1. | Data Display Numbering | |
| | | 10.9.2. | Mock Example Shell Referencing | |
| | | 10.9.3. | Deliverables | |
| | | 10.9.4. | Study Population Tables | |
| | | 10.9.5. | Safety Tables | |
| | | 10.9.6. | Safety Figures | |
| | | 10.9.7. | Pharmacokinetic Tables | |
| | | 10.9.9. | ICH Listings | |
| | | 10.9.10. | Non-ICH Listings | 6/ |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the CSR for Protocol: 213054.

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

This is an open-label, single-sequence, multiple-dose, 3 cohort study.

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

| Version / Release Date | Summary of Changes |
|---|---|
| Final 1.0 / 2021-02-24 | |
| Final 2.0 / 2021-10-15 | <ul> <li>Add Enrolled population as "All participants who passed screening and entered the study " for the presentation of .disposition analysis (Data display 1.1).</li> <li>In Section 5.2, change baseline for Cohort 3 Period 2 to Day 1 (Pre-Dose).</li> </ul> |

# 2.2. Study Objective(s) and Endpoint(s)

| | Objectives | Endpoints |
|---|---|---|
| | Primary | |
| Cohort 1 | To assess the effect of co-administration of DRV/ RTV 600/100 mg BID with GSK3640254 200 mg QD on the PK of GSK3640254 in healthy participants. | AUC(0-tau) and Cmax for<br>GSK3640254 |
| | To assess the effect of co-administration of<br>GSK3640254 200 mg QD with DRV/RTV<br>600/100 mg BID on the PK of DRV/RTV in<br>healthy participants. | AUC(0-tau), and Cmax for DRV/RTV |
| Cohort 2 | To assess the effect of co-administration of ETR 200 mg BID with GSK3640254 200 mg QD on the PK of GSK3640254 in healthy participants. To assess the effect of co-administration of | <ul> <li>AUC(0-tau) and Cmax for<br/>GSK3640254</li> <li>AUC(0-tau), and Cmax for ETR</li> </ul> |
| | ETR 200 mg BID with GSK3640254 200 mg QD on the PK of ETR in healthy participants. | |
| Cohort 3 | To assess the effect of co-administration of<br>ETR 200 mg BID and DRV/RTV 600/100 mg<br>BID with GSK3640254 200 mg QD on the PK<br>of GSK3640254 in healthy participants. | AUC(0-tau) and Cmax for<br>GSK3640254 |

| | Secondary |
|---|---|
| Cohort 1 | To assess the effect of co-administration of GSK3640254 200 mg QD with DRV/RTV 600/100 mg BID on the secondary PK parameters of DRV and RTV in healthy participants. Ctau, and Tmax for DRV, RTV, and GSK3640254 |
| Cohort 2 | To assess the effect of co-administration of GSK3640254 200 mg QD with ETR 200 mg BID on the secondary PK parameters of ETR in healthy participants. Ctau, and Tmax for ETR, and GSK3640254 GSK3640254 |
| Cohort 1, 2 & 3 | <ul> <li>To assess the safety and tolerability of GSK3640254 administered alone and in combination with DRV/RTV and/or ETR.</li> <li>Safety and tolerability endpoints include incidence of AEs, SAEs, AEs leading to discontinuation, deaths, marked laboratory abnormalities, and abnormalities in vital signs and 12-lead ECGs.</li> </ul> |

AE = adverse event; AUC(0-tau) = area under the plasma concentration-time curve from time zero to the end of the dosing interval at steady state; BID = twice daily; DRV = darunavir; Cmax = maximum observed concentration, Ctau = plasma concentration at the end of the dosing interval; ECG = electrocardiogram; ETR = etravirine; PK = pharmacokinetics; QD = once daily; RTV = ritonavir; SAE = serious adverse event; Tmax = time of maximum observed concentration.

### 2.3. Study Design



BID = twice daily; N = number of participants; QD = once daily.

# Design Features

A Phase 1, single-sequence, multiple-dose, 3 cohort study.

The study will consist of a screening period and a treatment period.

- Screening Period: within 28 days before the first dose of study intervention
- Treatment Period Cohort 1
  - Period 1: GSK3640254 200 mg tablets QD (Treatment A) on Days 1 through
     7.
  - Period 2: Darunavir (DRV)/ Ritonavir (RTV) 600/100 mg tablets twice daily (BID) (Treatment B) on Days 12 through 21.
  - Period 3: GSK3640254 200 mg tablets once daily (QD) (Treatment A) and DRV/RTV 600/100 mg tablets BID (Treatment B) on Days 22 through 31.
- Treatment Period Cohort 2
  - Period 1: GSK3640254 200 mg tablets QD (Treatment A) on Days 1 through
     7
  - Period 2: Etravirine (ETR) 200 mg tablets BID (Treatment C) on Days 12 through 21.
  - Period 3: GSK3640254 200 mg tablets QD (Treatment A) and ETR 200 mg tablets BID (Treatment C) on Days 22 through 31.
- Treatment Period Cohort 3
  - Period 1: GSK3640254 200 mg tablets QD (Treatment A) on Days 1 through
     7.
  - Period 2: GSK3640254 200 mg tablets QD (Treatment A), DRV/RTV 600/100 mg tablets BID (Treatment B), and ETR 200 mg tablets BID

| Overview of St | udy Design and Key Features |
|---|---|
| | (Treatment C) on Days 8 through 21. Per cohort, approximately 16 participants will be treated to ensure that 14 evaluable participants complete the study. |
| Dosing | <ul> <li>Treatment A: GSK3640254 200 mg tablets QD</li> <li>Treatment B: DRV/RTV 600/100 mg tablets BID</li> <li>Treatment C: ETR 200 mg tablets BID</li> </ul> |
| Time & Events | Refer to Appendix 1: Schedule of Activities |
| Treatment<br>Assignment | <ul> <li>PPD Clinical Pharmacology will remain open—label throughout the study. First 16 participants will be assigned to Cohort 3, and remaining 32 participants will be randomly assigned to Cohort 1 or 2.</li> </ul> |
| Interim<br>Analysis | No interim analysis is planned for this study |

# 2.4. Statistical Hypotheses

There is no formal hypothesis that will be statistically tested in this study.

Administration of GSK3640254 may change the exposure to DRV/RT and ETR, and administration of DRV/RTV and ETR may change the exposure to GSK3640254.

# 2.5. Sample Size Determination

As there is no formal research hypothesis being statistically tested in this study, the sample size was not selected based on statistical considerations but determined using feasibility. Per cohort, approximately 16 participants will be enrolled to ensure that 14 evaluable participants complete the study. If participants prematurely discontinue the study, additional participants may be enrolled after consultation with the sponsor to ensure that the required number of evaluable participants complete the study.

# 3. PLANNED ANALYSES

# 3.1. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) have been declared by Data Management.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who signed the informed consent form. | Study Population |
| Enrolled | All participants who passed screening and entered the study | Disposition |
| Randomized | All participants who are randomly assigned to a cohort. | Disposition |
| Safety | The Safety Population will include all participants who receive at least 1 dose of study medication. Participants will be analyzed according to the intervention they actually received. | <ul><li>Demographic</li><li>Safety</li></ul> |
| Pharmacokinetic<br>Concentration | The PK Concentration Population will include all participants who undergo plasma PK sampling and have evaluable PK assay results. | PK Concentration |
| Pharmacokinetic<br>Parameter | The PK Parameter Population will include all participants who undergo plasma PK sampling and have at least 1 evaluable PK parameter estimated. | <ul><li>PK Parameter</li><li>PK statistical<br/>analysis</li></ul> |

Refer to Appendix 9: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, participant management, or participant assessment) will be summarized and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Study Deviation Tool and Rules. The "significant" protocol deviation in the Study Deviation Tool and Rules is equivalent to "important" protocol deviations.

- Data will be reviewed prior to freezing the database to ensure all significant deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the electronic case record form (eCRF).

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| Data Displays for Reporting | | | |
| Description | Code | Order in TLF | Cohort Used |
| GSK3640254 200 mg tablets QD on Days 1 through 7. | Treatment A | 1 | Cohorts 1, 2, 3 |
| DRV/RTV 600/100 mg tablets twice daily (BID) (Treatment B) on Days 12 through 21. | Treatment B | 2 | Cohort 1 |
| GSK3640254 200 mg tablets QD and DRV/RTV 600/100 mg tablets BID on Days 22 through 31. | Treatment A + Treatment B | 3 | Cohort 1 |
| ETR 200 mg tablets BID on Days 12 through 21. | Treatment C | 4 | Cohort 2 |
| GSK3640254 200 mg tablets QD and ETR 200 mg tablets BID on Days 22 through 31. | Treatment A + Treatment C | 5 | Cohort 2 |
| GSK3640254 200 mg tablets QD, DRV/RTV 600/100 mg tablets BID, and ETR 200 mg tablets BID on Days 8 through 21. | Treatment A + Treatment B +Treatment C | 6 | Cohort 3 |

# 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions), baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.

#### Cohorts 1 and 2:

| Parameter | Study Assessments Considered as Baseline | | | | | Baseline | Used in Data | a Display |
|---|---|---|---|---|---|---|---|---|
| | Check-in Baseline Day 1 Day 12 Day 22 (Pre-dose) (Pre-dose) | | Period 1 | Period 2 | Period 3 &<br>Follow-up | | | |
| Vital Sign | X | X | X | Х | Х | Day 1<br>(Pre-Dose) <sup>[1]</sup> | Day 12<br>(Pre-Dose) <sup>[1]</sup> | Day 22<br>(Pre-Dose) <sup>[1]</sup> |
| 12-Lead<br>ECG | Х | Х | Х | Х | Х | Day 1<br>(Pre-Dose) <sup>[1]</sup> | Day 12<br>(Pre-Dose) <sup>[1]</sup> | Day 22<br>(Pre-Dose) <sup>[1]</sup> |

<sup>[1]</sup> The average (for blood pressure, pulse, and ECG numeric assessment) or the worst case (for ECG interpretation - Normal> Abnormal, Not Clinical Significant> Abnormal, Clinically Significant) of the pre-dose triplicate assessments will be used as the baseline.

#### Cohort 3:

| Parameter | Study Asse | essments C | onsidered as I | Baseline Used<br>Display | in Data | |
|---|---|---|---|---|---|---|
| | Check-in Baseline Day 1 Day 8 (Pre-dose) | | Period 1 | Period 2 and follow-up | | |
| Vital Sign | Х | Х | Х | Х | Day 1<br>(Pre-Dose) <sup>[1]</sup> | Day 8<br>(Pre-Dose) <sup>[1]</sup> |
| 12-Lead<br>ECG | Х | Х | Х | Х | Day 1<br>(Pre-Dose) <sup>[1]</sup> | Day 1<br>(Pre-Dose) <sup>[1]</sup> |

<sup>[1]</sup> The average (for blood pressure, pulse, and ECG numeric assessment) or the worst case (for ECG interpretation - Normal> Abnormal, Not Clinical Significant> Abnormal, Clinically Significant)) of the pre-dose triplicate assessments will be used as the baseline

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Schedule of Activities |
| 10.2 | Appendix 2: Study Phase and Treatment Emergent Adverse Event |
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Reporting Standards for Missing Data |
| 10.6 | Appendix 6: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events |
| 10.7 | Appendix 7: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "Safety", "Randomized" or "Screened", population, unless otherwise specified.

Study population analyses including analyses of participant's disposition, protocol deviations (including inclusion/exclusion criteria deviations), demographic and baseline characteristics, prior and concomitant medications, and exposure will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 9: List of Data Displays.

#### 7. PHARMACOKINETIC ANALYSES

### 7.1. Primary Pharmacokinetic Analyses

#### 7.1.1. Endpoint / Variables

#### 7.1.1.1. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Standards for PK). Plasma concentrations of GSK3640254, DRV, RTV, and ETR will be measured and presented in tabular form and will be summarized descriptively. Plasma GSK3640254, DRV, RTV, and ETR concentration-time data will be listed by participant, treatment group, and sampling time and summarized by treatment group and sampling time.

#### 7.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin (8.0 or higher). All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits. Subjects who experience emesis at or before 2 times median  $T_{max}$  for the given treatment will be excluded from the calculation of summary statistics and statistical analysis for the respective treatment.

| Parameter | Parameter Description |
|---|---|
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| AUC(0-tau) | Area under the plasma concentration-time curve from time 0 to the end of the dosing interval at steady state, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| NOTES: | |
| <ul> <li>Additional</li> </ul> | parameters may be included as required. |

# 7.1.2. Summary Measure

Pharmacokinetic parameters AUC(0-tau) and Cmax following administration of GSK3640254 with or without administration of DRV/RTV and/or ETR to healthy participants.

#### 7.1.3. Population of Interest

The primary PK analyses will be based on the PK concentration population for plasma PK concentrations and the PK parameter population for plasma PK parameters and statistical analysis.

### 7.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarized using descriptive statistics, graphically presented (where appropriate), and listed

Primary plasma PK parameters (AUC[0-tau] and Cmax) will be estimated for GSK3640254, DRV, RTV, and ETR. Summary statistics (arithmetic mean, geometric mean, median, standard deviation [SD], minimum, maximum, between-subject coefficient of variation [CVb], and 95% CI for plasma PK parameter values) will be summarized by treatment.

#### 7.1.4.1. Statistical Methodology Specification

The following PK statistical analyses will only be performed if sufficient data are available (i.e. if participants have well defined plasma profiles).

#### **Endpoint / Variables**

Plasma primary PK endpoints include AUC(0-tau) and Cmax, as data permit

#### **Model Specification**

- Analysis will be performed to compare the PK exposure of GSK3640254 with and
  without DRV/RTV (Cohort 1), ETR (Cohort 2), or DRV/RTV/ETR (Cohort 3). Analyses will be performed
  on the natural logarithms of AUC(0-tau) and Cmax using linear mixed-effect models with treatment as a
  fixed effect, and measurements within participant as repeated measures, and subject as a random
  effect.
- Effects will be estimated, and CIs will be constructed for the following treatment comparisons:

Treatment A+B versus Treatment A (Cohort 1)

Treatment A+C versus Treatment A (Cohort 2)

Treatment A+B+C versus Treatment A (Cohort 3)

- Point estimates and 90% CIs for treatment differences on the log scale derived from the model will be exponentiated to obtain estimates for geometric mean ratios and CIs on the original scale.
- Analysis will be performed to compare the PK exposure of DRV (Cohort 1), RTV (Cohort 1), and ETR (Cohort 2) with and without GSK3640254. Analyses will be performed on the natural logarithms of AUC(0-tau) and Cmax using linear mixed-effect models with treatment as a fixed effect, and measurements within participant as repeated measures, and subject as a random effect.
- Effects will be estimated, and CIs will be constructed for the following treatment comparisons: Treatment A+B versus Treatment B (Cohort 1)
  - Treatment A+C versus Treatment C (Cohort 2)
- Point estimates and 90% CIs for treatment differences on the log scale derived from the model will be exponentiated to obtain estimates for geometric mean ratios and CIs on the original scale.

#### **Model Checking & Diagnostics**

Model assumptions will be applied, but appropriate adjustments may be made based on the data.

#### **Model Results Presentation**

• Statistical analysis by analysis of variance (ANOVA) will be presented in tabular format with geometric mean ratios and 90% CIs for:

Treatment A+B versus Treatment A (Cohort 1)

Treatment A+C versus Treatment A (Cohort 2)

Treatment A+B+C versus Treatment A (Cohort 3)

 Statistical analysis by analysis of variance (ANOVA) will be presented in tabular format with geometric mean ratios and 90% CIs for:

Treatment A+B versus Treatment B (Cohort 1)

Treatment A+C versus Treatment C (Cohort 2)

#### 7.2. Secondary Pharmacokinetic Analyses

#### 7.2.1. Endpoint / Variables

#### 7.2.1.1. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Standards for PK)

#### 7.2.1.2. Derived Pharmacokinetic Parameters

Plasma PK parameters listed below will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|-----------|--------------------------------------------------------|
| Tmax | Time of maximum observed concentration |
| Ctau | Plasma concentration at the end of the dosing interval |

#### NOTES:

Additional parameters may be included as required.

If additional pharmacokinetic parameters are needed they will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin (8.0 or higher). All calculations of non-compartmental parameters will be based on actual sampling times. Subjects who experience emesis at or before 2 times median  $T_{max}$  for the given treatment will be excluded from the calculation of summary statistics and statistical analysis for the respective treatment.

#### 7.2.2. Summary Measure

Pharmacokinetic parameters Tmax and Ctau of GSK3640254, DRV, RTV, and ETR following administration of GSK3640254 with or without administration of DRV/RTV and/or ETR to healthy participants.

#### 7.2.3. Population of Interest

The secondary PK analyses will be based on the PK concentration population for plasma PK concentrations, and the PK parameter population for plasma and statistical analysis, unless otherwise specified.

#### 7.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 7.1.1 will be summarized using descriptive statistics, graphically presented (where appropriate), and listed.

Secondary plasma PK parameters (Tmax and Ctau) will be estimated for GSK3640254, DRV, RTV and ETR. Summary statistics (arithmetic mean, geometric mean, median, SD, minimum, maximum, and coefficient of variation) for plasma PK parameter values will be summarized by treatment.

Additionally, pre-dose (trough) PK plasma concentrations of GSK3640254, DRV, RTV, and ETR will be summarized and used to assess achievement of steady state.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population unless otherwise specified.

#### 8.1. Adverse Events Analyses

Adverse events (AEs) analyses including the analysis of AEs, serious AEs (SAEs), AEs of special interest (AESI), and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 9: List of Data Displays.

For studies with greater than one treatment period (e.g., crossover study), if AE onset is during one period and worsens during a later period, it will be counted in both periods. For the later period the onset date of AE with the elevated grade will be the first dose date of the later treatment period.

#### 8.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of chemistry laboratory tests, hematology laboratory tests, urinalysis, liver function tests, and pregnancy test will be based on GSK Core Data Standards and will be graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (Version 2.1, July 2017). The details of the planned displays are in Appendix 9: List of Data Displays.

#### 8.3. Adverse Events of Special Interest

At the end of the study, QT prolongation, gastrointestinal intolerability, gastric toxicity, psychiatric events, nervous system disorders, and skin and subcutaneous tissue disorders will be summarized by treatment. A listing will also be provided accordingly.

The AESI of QT prolongation will be defined as cardiac disorders system organ class (SOC) plus preferred terms (PTs) using the Medical Dictionary for Regulatory Activities (MedDRA) Standardized MedDRA Query (SMQ) "Torsade de pointes/QT Prolongation" (narrow and broad terms) plus seizure.

Gastrointestinal intolerability and gastric toxicity AESIs will be defined within three narrow sub-SMQs [Gastrointestinal nonspecific symptoms and therapeutic procedures SMQ; Gastrointestinal nonspecific dysfunction SMQ; Gastrointestinal nonspecific inflammation (SMQ)] plus a selection of relevant broad PTs from the Gastrointestinal non-specific symptoms and therapeutic procedures SMQ.

Psychiatric AESI will be defined within the following:

- Sub-SMQ "Suicide/self-injury" (SMQ) from parent SMQ of "Depression and Suicide/Self Injury". Only narrow terms from the sub-SMQ will be selected.
- Sub-SMQ "Depression (excluding suicide and self-injury)" (SMQ) from parent SMQ of "Depression and Suicide/Self Injury". Only narrow terms from the sub-SMQ will be selected.

- All PTs from high level group term (HLGT) "Manic and Bipolar Mood Disorders and Disturbances" under SOC "Psychiatric Disorders".
- Narrow terms from SMQ "Psychosis and Psychotic Disorders" selected.
- All PTs from HLGT "Anxiety Disorders and Symptoms", under SOC "Psychiatric disorders".
- All PTs from HLGT "Sleep Disorders and Disturbances" and HLGT "Sleep disturbances (include subtypes)".

Nervous system disorders AESIs will be defined within the following:

• Four HLGTs under Nervous System Disorders SOC: "Headaches"; "Mental impairment disorders (excluding dementia)"; "Disturbance in consciousness" and "Seizures and seizure disorder"

Skin and subcutaneous tissue disorder AESIs will be defined with the following PTs:

Dermatitis, Dermatitis allergic, Dermatitis atopic, Eczema, Eczema eyelids, Eczema nummular, Eyelid irritation, Skin irritation, Urticarial dermatitis, Eyelid pruritis, Pruritus, Pruritus allergic, Rash pruritic, Rash, Rash macular, Rash maculopapular, Rash morbilliform, Rash papular, Rash pruritic, Urticaria, Drug eruption and Rash pustular

### 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs, vital signs, liver events, and Columbia Suicide Severity Rating Scale (C-SSRS) will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 9: List of Data Displays.

# 8.5. COVID 19 Related Analyses

Based on GSK's "Impact of COVID-19 on Assessment of Safety in Clinical Trials Points to Consider", it is GSK's recommendation that study teams should capture COVID-19 cases based on the WHO criteria using the categories of: suspected, probable, and confirmed cases. COVID-19 eCRF pages are used in the study for data collection and analysis purposes. After a discussion with the study team, the following analyses will be included:

- Number of subjects with suspected, probable, or confirmed COVID-19 infection
- Number of subjects who had a COVID-19 diagnosis test performed and the number of subjects with positive, negative, or indeterminate results
- Incidence of COVID-19 as reported as an AE and SAE
- Incidence of treatment discontinuation due to an AE of COVID-19 infection
- Severity, duration, and outcome of COVID-19 AEs

If percentage of COVID-19 cases is >10% (> 5 subjects with an AE of COVID-19), a summary of COVID-19 symptoms for subjects with COVID-19 AE will be added.

Further display details are provided in Appendix 9: List of Data Displays.

# 9. REFERENCES

ViiV Healthcare group of companies Document Number 2020N432810\_00 (10SEP2020) Open-Label, Single-Sequence Study to Evaluate the Effects of Darunavir/Ritonavir and/or Etravirine on the Pharmacokinetics of GSK3640254 and the Effects of GSK3640254 on the Pharmacokinetics of Darunavir/Ritonavir and/or Etravirine in Heathy Adults

# 10. APPENDICES

# 10.1. Appendix 1: Schedule of Activities

#### 10.1.1. Protocol Defined Schedule of Events

# **Screening Visit**

| Procedure | Screening<br>(up to 28 days before Day 1) |
|---|---|
| Outpatient visit | X |
| Informed consent | X |
| Inclusion and exclusion criteria | X |
| Demography | X |
| Full physical examination including height and weight <sup>0</sup> | X |
| Laboratory assessments (hematology, clinical chemistry, urinalysis) | X |
| 12-lead electrocardiogram | X |
| Vital sign measurements | X |
| Medication/drug/alcohol history | X |
| Past and current medical conditions | X |
| Columbia-Suicide Severity Rating Scale | X |
| Serum pregnancy test | X |
| Follicle-stimulating hormone (as needed, to confirm postmenopausal status) | X |
| Drug, alcohol, and cotinine screen | X |
| Human immunodeficiency virus, Hepatitis B and C screening | X |
| Molecular test for SARS-CoV-2b | |

a. A full physical examination will include at a minimum, assessments of the skin, cardiovascular, respiratory, gastrointestinal, and neurological systems.

b. Two consecutive approved molecular tests (polymerase chain reaction or antigen test). The first test should be performed ≥7 days prior to admission.

# **Time and Events Table - Cohort 1**

| Procedure | Check-<br>in | Baseline | 1 | P<br>Freatmer<br>Washou | | ays 1-7 | ) | Perio<br>Treatm<br>(Days | nent B | | | Treatme | | Period 3 reatmen | | ys 22-3 | 31) | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day -1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8-10 | Day<br>11 | Days<br>12-20 | Day<br>21 | Day<br>22 | Day<br>23 | Days 24-25 | Day<br>26 | Days<br>27-30 | Day<br>31 | Day<br>32 | Days<br>33-34 | Day<br>35 | |
| Admit to clinic | Χ | | | | | | | | | | | | | | | | | | |
| Discharge from clinic | | | | | | | | | | | | | | | | | | Х | |
| Brief physical examination | Х | | | | х | | Х | | х | | | | х | | | | | х | Includes, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). |
| Vital sign<br>measurements | Х | X | X | D2 | X | | Х | D12,<br>D13,<br>D17 | | Х | X | | X | | | | | X | Blood pressure<br>and pulse<br>measured in<br>triplicate at<br>pre-dose on Days<br>1, 12, and 22.<br>Single blood<br>pressure and<br>pulse will be<br>measured on other<br>study days. |
| Temperature<br>Check | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | |

| Procedure | Check-<br>in | Baseline | 7 | P<br>reatmer<br>Washou | | ays 1-7 | ) | Perio<br>Treatm<br>(Days 1 | ent B | | | Treatme | | Period 3<br>reatmen | | ys 22-3 | 1) | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day –1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8-10 | Day<br>11 | Days<br>12-20 | Day<br>21 | Day<br>22 | Day<br>23 | Days<br>24-25 | Day<br>26 | Days<br>27-30 | Day<br>31 | Day<br>32 | Days<br>33-34 | Day<br>35 | |
| 12-lead ECG | X | | X | | X | | X | D12 | X | X | | | X | | | | | X | ECGs on Days 1,<br>12, and 22, will be<br>taken pre-dose,<br>and at 2 and 4 and<br>6 hours post-dose.<br>Pre-dose ECGs on<br>Days 1, 12, and 22<br>will be taken in<br>triplicate. The<br>post-dose ECGs<br>are single ECGs. |
| Drug, alcohol,<br>and cotinine<br>screen | Х | | | | | | | | | | | | | | | | | | See Protocol<br>Appendix 2 for<br>tests. |
| Laboratory<br>assessments<br>(hematology,<br>clinical<br>chemistry,<br>urinalysis) | Х | | | | Х | | Х | | Х | | | | Х | | | | | Х | See Protocol<br>Appendix 2 for<br>tests. |

| Procedure | Check-<br>in | Baseline | | P<br>reatmer<br>Washou | | ays 1-7 | ) | Perio<br>Treatm<br>(Days | ent B | | 7 | Freatme | | Period 3<br>reatmen | | ys 22-3 | 1) | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day -1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8-10 | Day<br>11 | Days<br>12-20 | Day<br>21 | Day<br>22 | Day<br>23 | Days<br>24-25 | Day<br>26 | Days<br>27-30 | Day<br>31 | Day<br>32 | Days<br>33-34 | Day<br>35 | |
| Molecular test<br>for SARS-CoV | X1 | | | D6 | | | | D13,<br>D20 | | | | | | D27 | | | | X | Test to be obtained every 7 days from Checkin (regardless of period or washout) while in-house. ¹The second test should be performed 24 hours prior to admission to the unit. Participants should be quarantined within the unit until the second test result is negative. Once the second test result is confirmed to be negative, they can be released into the unit and follow infection control practices. |
| Pregnancy<br>test | X | | | | | | | | | | | | | | | | | Χ | Urine pregnancy test to confirm status. |
| Columbia-<br>Suicide | Х | | | | | | Х | | | Х | | | | | Х | | | | See Protocol<br>Section 8.2.6 for |

| Procedure | Check-<br>in | Baseline | - | P<br>Treatmer<br>Washor | | ays 1-7 | | Perio<br>Treatm<br>(Days | nent B | | | Treatme | | Period 3<br>reatmen | | ys 22-3 | 31) | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day –1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8-10 | Day<br>11 | Days<br>12-20 | Day<br>21 | Day<br>22 | Day<br>23 | Days 24-25 | Day<br>26 | Days 27-30 | Day<br>31 | Day<br>32 | Days<br>33-34 | Day<br>35 | |
| Severity<br>Rating Scale | | | | | | | | | | | | | | | | | | | details. |
| Study<br>intervention:<br>DRV/RTV<br>(BID) | | | | | | | | Х | Х | Х | Х | X | Х | X | Х | | | | See Protocol<br>Section 6.1 for<br>study intervention<br>details. |
| Study<br>intervention:<br>GSK3640254<br>200 mg (QD) | | | Х | Х | Х | | | | | Х | X | X. | Х | X | Х | | | | See Protocol<br>Section 6.1 for<br>study intervention<br>details. |
| DRV/RTV PK sampling | | | | | | | | D19,<br>D20 | X | | | | | | X | | | | Pre-dose Days 19, 20 and 21. Post Day 21 dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose. Pre-dose Day 31. Post Day 31 dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours. |
| GSK3640254<br>PK sampling | | | | D5,<br>D6 | X | D8 | | | | | | | | D29,<br>D30 | Х | X | | | Pre-dose Days 5,<br>6, and 7. Post<br>Day 7 dose at 0.5,<br>1, 1.5, 2, 3, 4, 6,<br>8, 12, 16, and<br>24 hours.<br>Pre-dose Days<br>29, 30, and 31. |

| Procedure | Check-<br>in | Baseline | | P<br>Treatme<br>Washo | | ays 1-7 | | Perio<br>Treatm<br>(Days | ent B | | | Treatme | | Period 3 reatmen | | ys 22-3 | 1) | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day –1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8-10 | Day<br>11 | Days<br>12-20 | Day<br>21 | Day<br>22 | Day<br>23 | Days<br>24-25 | Day<br>26 | Days<br>27-30 | Day<br>31 | Day<br>32 | Days<br>33-34 | Day<br>35 | |
| | | | | | | | | | | | | | | | | | | | Post Day 31 dose<br>at 0.5, 1, 1.5, 2, 3,<br>4, 6, 8, 12, 16,<br>and 24 hours. |
| AE review | | | + | -==== | ===== | ===== | | ====== | | ===== | ===== | | ===== | | ===== | ===== | | $\rightarrow$ | |
| SAE review | | • | -==== | | ===== | | | ===== | | | ===== | | ===== | | | ===== | | ===> | |
| Concomitant medication review | | • | -==== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===→ | |

Abbreviations: AE = adverse event; BID = twice daily; D = day; DRV = darunavir; ECG = electrocardiogram; PK = pharmacokinetic; QD = once daily; RTV = ritonavir; SAE = serious adverse event.

#### **Time and Events Table - Cohort 2**

| Procedure | Check-<br>in | Baseline | | P<br>reatmer<br>Washou | | ays 1- | | Perio<br>Treati<br>C<br>(Days | ment<br>;<br>; 12- | | 1 | Γreatme | nt A +1 | Period<br>reatme | | ays 22 | -31) | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day -1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8-<br>10 | Day<br>11 | Days<br>12-20 | Day<br>21 | Day<br>22 | Day<br>23 | Days<br>24-25 | Day<br>26 | Days<br>27-30 | Day<br>31 | Day<br>32 | Days<br>33-35 | Day<br>36 | |
| Admit to clinic | Х | | | | | | | | | | | | | | | | | | |
| Discharge from clinic | | | | | | | | | | | | | | | | | | Χ | |

| Procedure | Check-<br>in | Baseline | | P<br>reatmer<br>Washou | | ays 1 | | Perio<br>Treati<br>C<br>(Days | ment | | | Treatme | nt A +1 | Period<br>Freatmen | | ays 22 | -31) | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day -1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8-<br>10 | Day<br>11 | Days<br>12-20 | Day<br>21 | Day<br>22 | Day<br>23 | Days 24-25 | Day<br>26 | Days<br>27-30 | Day<br>31 | Day<br>32 | Days<br>33-35 | Day<br>36 | |
| Brief physical examination | Х | | | | Х | | X | | X | | | | X | | | | | Х | Includes, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). |
| Vital sign<br>measurements | Х | Х | X | D2 | X | | Х | D12,<br>D13,<br>D17 | | Х | Х | | Х | | | | | Х | Blood pressure and pulse measured in triplicate at pre-dose on Days 1, 12, and 22. Single blood pressure and pulse will be measured on other study days. |
| Temperature<br>Check | X | X | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | Х | Х | Х | Х | Х | Х | |

| Procedure | Check-<br>in | Baseline | | P<br>reatmer<br>Washou | | ays 1 | | Perio<br>Treate<br>(Days | ment<br>;<br>s 12- | | | Treatme | nt A + | Period<br>Treatme | | ays 22 | -31) | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day -1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8-<br>10 | Day<br>11 | Days<br>12-20 | Day<br>21 | Day<br>22 | Day<br>23 | Days 24-25 | Day<br>26 | Days 27-30 | Day<br>31 | Day<br>32 | Days<br>33-35 | Day<br>36 | |
| 12-lead ECG | Х | Х | Х | | Х | | Х | D12 | Х | X | | | X | | | | | Х | ECGs on Days 1, 12, and 22, will be taken predose, and at 2, 4, and 6 hours post-dose. Pre-dose ECGs on Days 1, 12, and 22 will be taken in triplicate. The post-dose ECGs are single ECGs. |
| Drug, alcohol,<br>and cotinine<br>screen | Х | | | | | | | | | | | | | | | | | | See Protocol Appendix 2 for tests. |
| Laboratory<br>assessments<br>(hematology,<br>clinical<br>chemistry,<br>urinalysis) | Х | | | | Х | | Х | | Х | | | | Х | | | | | Х | See Protocol Appendix 2 for tests. |

| Procedure | Check-<br>in | Baseline | | Period 1<br>Treatment A (Days 1-7)<br>Washout (Days 8-11) | | | | | Period 2 Treatment C (Days 12- 21) Period 3 Treatment A +Treatment C (Days 22-31) Period 3 Treatment A +Treatment C (Days 22-31) | | | | | | | | | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day -1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8-<br>10 | Day<br>11 | Days<br>12-20 | Day<br>21 | Day<br>22 | Day<br>23 | Days<br>24-25 | Day<br>26 | Days 27-30 | Day<br>31 | Day<br>32 | Days<br>33-35 | Day<br>36 | |
| Molecular test<br>for<br>SARS-CoV-2 | X1 | | | D6 | | | | D13,<br>D20 | | | | | | D27 | | | | X | Test to be obtained every 7 days from Check-in (regardless of period or washout) while in-house. ¹The second test should be performed 24 hours prior to admission to the unit. Participants should be quarantined within the unit until the second test result is negative. Once the second test result is confirmed to be negative, they can be released into the unit and follow infection control practices. |
| Pregnancy test | Х | | | | | | | | | | | | | | | | | Х | Urine pregnancy test to confirm status. |
| Columbia-<br>Suicide<br>Severity<br>Rating Scale | Х | | | | | | х | | | Х | | | | | Х | | | | See Protocol Section<br>8.2.6 for details. |
| Study intervention: ETR (BID) | | | | | | | | Х | Х | Х | Х | Х | Х | Х | Х | | | | See Protocol Section<br>6.1 for study<br>intervention details. |

| Procedure | Check-<br>in | Baseline | | Period 1<br>Treatment A (Days 1-7)<br>Washout (Days 8-11) | | | | | Period 2 Treatment C (Days 12- 21) Period 3 Treatment A +Treatment C (Days 22-31) Period 3 Treatment A +Treatment C (Days 22-31) | | | | | | | | | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day -1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8-<br>10 | Day<br>11 | Days<br>12-20 | Day<br>21 | Day<br>22 | Day<br>23 | Days<br>24-25 | Day<br>26 | Days 27-30 | Day<br>31 | Day<br>32 | Days<br>33-35 | Day<br>36 | |
| Study<br>intervention:<br>GSK3640254<br>200 mg (QD) | | | Х | Х | Х | | | | | Х | Х | X. | Х | Х | Х | | | | See Protocol Section<br>6.1 for study<br>intervention details. |
| ETR PK sampling | | | | | | | | D19,<br>D20 | X | | | | | | Х | | | | Pre-dose Days 19, 20<br>and 21. Post Day 21<br>dose at 0.5, 1, 1.5, 2, 3,<br>4, 6, 8, and 12 hours<br>post-dose.<br>Pre-dose Day 31. Post<br>Day 31 dose at 0.5, 1,<br>1.5, 2, 3, 4, 6, 8, and<br>12 hours. |
| GSK3640254<br>PK sampling | | | | D5,<br>D6 | Х | D8 | | | | | | | | D29,<br>D30 | Х | Х | | | Pre-dose Days 5, 6, and 7. Post Day 7 dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours. Pre-dose Days 29, 30, and 31. Post Day 31 dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours. |
| AE review | | | <b>←==</b> | ===== | | | | ===== | | | ===== | | | ===== | | | ===== | ===→ | |
| SAE review | | <b>←====</b> | | | ===== | ==== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ====== | ===== | | ===== | ===→ | |


213054

| Procedure | Check-<br>in | Baseline | | P<br>reatmer<br>Washor | | ays 1- | | Perio<br>Treati<br>C<br>(Days | ment<br>;<br>s 12- | | - | <b>Freatme</b> | nt A +1 | Period<br>Freatme | | ays 22 | -31) | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day -1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8-<br>10 | Day<br>11 | Days<br>12-20 | Day<br>21 | Day<br>22 | Day<br>23 | Days 24-25 | Day<br>26 | Days<br>27-30 | Day<br>31 | Day<br>32 | Days<br>33-35 | Day<br>36 | |
| Concomitant medication review | | <b>←===</b> = | ==== | ===== | ==== | ===== | ===== | ===== | ===== | ===== | ==== | ===== | ==== | ===== | ===== | ==== | ===== | ===> | |

Abbreviations: AE = adverse event; BID = twice daily; D = day; ECG = electrocardiogram; ETR = etravirine; PK = pharmacokinetic; QD = once daily; SAE = serious adverse event.

# **Time and Events Table - Cohort 3**

| Procedure | Check- | Baseline | Tr | Period 1<br>eatment<br>Days 1-7 | Α | | | Tre | | Notes | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day -1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8 | Day<br>9 | Days<br>10-12 | Day<br>13 | Day<br>14 | Days<br>15-16 | Day<br>17 | Days<br>18-20 | Day<br>21 | Day<br>22 | Days<br>23-25 | Day<br>26 | |
| Admit to clinic | Χ | | | | | | | | | | | | | | | | | |
| Discharge from clinic | | | | | | | | | | | | | | | | | Х | |
| Brief physical examination | х | | | | х | | | | | Х | | | | | | | Х | Includes, at a minimum,<br>assessments of the skin, lungs,<br>cardiovascular system, and abdomen<br>(liver and spleen). |
| Vital sign<br>measurements | х | Х | Х | D2 | Х | Х | | | | Х | | Х | | | | | Х | Blood pressure and pulse measured in triplicate at pre-dose on Days 1 and 8. Single blood pressure and pulse will be measured on other study days. |
| Temperature<br>Check | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | |
| 12-lead ECG | х | Х | Х | | | Х | Х | | | | | | | | | | Х | ECGs on Days 1, 8, and 9 will be taken pre-dose, and at 2, 4, and 6 hours post-dose. Pre-dose ECGs on Days 1, 8, and 9 will be taken in triplicate. The post-dose ECGs are single ECGs. |
| Drug, alcohol,<br>and cotinine<br>screen | Х | | | | | | | | | | | | | | | | | See Protocol Appendix 2 for tests. |

| Procedure | | | | | | | | Tre | | Notes | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day -1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8 | Day<br>9 | Days<br>10-12 | Day<br>13 | Day<br>14 | Days<br>15-16 | Day<br>17 | Days<br>18-20 | Day<br>21 | Day<br>22 | Days<br>23-25 | Day<br>26 | |
| Laboratory<br>assessments<br>(hematology,<br>clinical<br>chemistry,<br>urinalysis) | х | | | | X | | | | | х | | | | | | | Х | See Protocol Appendix 2 for tests. |
| Molecular Test<br>for SARS-CoV-<br>2 | X <sup>1</sup> | | | D6 | | | | | х | | | | D20 | | | | Х | Test to be obtained every 7 days from Check-in (regardless of period or washout) while in-house. 1 The second test should be performed 24 hours prior to admission to the unit. Participants should be quarantined within the unit until the second test result is negative. Once the second test result is confirmed to be negative, they can be released into the unit and follow infection control practices. |
| Pregnancy test | Х | | | | | | | | | | | | | | | | Х | Urine pregnancy test to confirm status. |
| Columbia-<br>Suicide<br>Severity Rating<br>Scale | Х | | | | | х | | | х | | | | | Х | | | | See Protocol Section 8.2.6 for details. |
| Study<br>intervention:<br>DRV/RTV and<br>ETR (BID) | | | | | | х | X | Х | х | х | х | Х | х | х | | | | See Protocol Section 6.1 for study intervention details. |

| Procedure | Check-<br>in | Baseline | Tr | Period 1<br>Treatment A<br>(Days 1-7) | | | Treatment A + Treatment B + Treatment C (Days 8-21) | | | | | | | | | | | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –2 | Day -1 | Day<br>1 | Days<br>2-6 | Day<br>7 | Day<br>8 | Day<br>9 | Days<br>10-12 | Day<br>13 | Day<br>14 | Days<br>15-16 | Day<br>17 | Days<br>18-20 | Day<br>21 | Day<br>22 | Days<br>23-25 | Day<br>26 | | |
| Study<br>intervention:<br>GSK3640254<br>200 mg (QD) | | | х | Х | Х | Х | Х | Х | Х | Х | X. | Х | Х | х | | | | See Protocol Section 6.1 for study intervention details. | |
| DRV/RTV and<br>ETR PK<br>sampling | | | | | | | | | | | | | D19,<br>D20 | Х | | | | Pre-dose Days 19, 20, and 21. Post<br>Day 21 dose at 0.5, 1, 1.5, 2, 3, 4, 6,<br>8, and 12 hours. | |
| GSK3640254<br>PK sampling | | | | D5,<br>D6 | Х | Х | | | | | | | | х | Х | | | Pre-dose Days 5, 6, and 7. Post Day 7 dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours. Pre-dose Day 21. Post Day 21 dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours. | |
| AE review | | | | <del>(</del> ===== | ===== | ===== | ====== | ====== | ===== | ===== | ====== | ===== | ====== | ===== | ===== | ======- | <del>)</del> | | |
| SAE review | | <b>←</b> = | ===== | ====== | | | ====== | ====== | ===== | ===== | ====== | ===== | ====== | ===== | ===== | ====== | <del>)</del> | | |
| Concomitant medication review | | <b>←</b> = | ===== | ===== | | | | | | | | | ===== | | | | | thu DTV - site and in CAF - and an | |

AE = adverse event; BID = twice daily; D = day; DRV = darunavir; ECG = electrocardiogram; ETR = etravirine; PK = pharmacokinetic; QD = once daily; RTV = ritonavir; SAE = serious adverse event.

• Participants will fast overnight for at least 8 hours prior to breakfast and before the AM dose and for at least 2 hours prior to dinner and before the PM dose. Participants will receive the moderate fat meal 30 minutes prior to dosing. Participants will eat this meal in 25 minutes or less. Dose administration will occur within 5 minutes of completion of meal consumption.

- Serial PK blood samples will be collected before (at 0 hour) and after the AM study drug administration at the time points listed. For the study interventions that are administered twice daily (BID) (DRV/RTV and ETR), the 12-hour sample will be collected before the PM dose.
- Day 35 for Cohort 1, Day 36 for Cohort 2, and Day 26 for Cohort 3 is study discharge. Evaluations scheduled for study discharge will also be performed for participants who discontinue prior to completing.
- The timing of planned study assessments may change during the course of the study based on emerging data/in-stream data review (e.g., to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.

Any changes in the timing of time points for any planned study assessments as the result of emerging PK data from this study must be documented and approved by the relevant study team member and then archived in the sponsor and site study files but will not constitute a protocol amendment. The Institutional Review Board/ Independent Ethics Committee will be informed of any safety issues that constitute a substantial amendment and require alteration of the safety monitoring scheme or amendment of the informed consent form. The changes will be approved by the health authority and the ethics committee before implementation

# 10.2. Appendix 2: Study Phases and Treatment Emergent Adverse Events

# 10.2.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment start date(/time) and stop date(/time).

#### 10.2.1.1. Study Phases for Lab, Electrocardiograms, and Vital Signs

Assessments and events will be classified according to the time of occurrence relative to study treatment start date(/time) and stop date(/time).

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date and Time ≤Study Treatment Start Date and Time |
| On-Treatment | Study Treatment Start Date and Time <date +="" 5="" and="" date="" days<="" stop="" td="" time="" treatment="" ≤study=""></date> |
| Post-Treatment | Date and Time >Study Treatment Stop Date and Time + 5 days |

#### 10.2.1.2. Study Phases for Concomitant Medication

| Study Phase | Study Phase |
|-------------|-------------|
| Prior | Prior |
| Concomitant | Concomitant |

#### **NOTES:**

Please refer to Appendix 5: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 10.2.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>If AE onset date and time is on or after treatment start date and time &amp; on or before treatment stop date and time + 5 days.</li> <li>Study Treatment Start Date and Time ≤AE Start Date and Time ≤Study Treatment Stop Date and Time + 5 days.</li> <li>If the AE onset date is completely missing, the AE is considered as treatment emergent.</li> </ul> |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Please refer to Appendix 5: Reporting Standards for Missing Data for handling of missing and partial dates for AEs. Use the rules in this table if the AE onset date is completely missing.

#### 10.3. Appendix 3: Data Display Standards & Handling Conventions

#### 10.3.1. **Reporting Process**

| Software | |
|-------------------|-----------------------------------------------------|
| The currently sup | ported versions of SAS software (9.4) will be used. |
| Reporting Area | |
| HARP Server | \\us1salx00259.corpnet2.com |
| HARP Compound | \gsk3640254\mid213054\final_01 |
| Analysis Datasets | |

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.1).
- For creation of ADaM datasets (ADC1/ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for all reporting efforts described in the RAP.

#### 10.3.2. Reporting Standards

#### General

The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK Clinical Study Report. All participant level listings should be located in the modular appendices as ICH or non-ICH listings.

#### **Formats**

- All data will be reported according to the actual treatment the participant received unless otherwise
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be rounded to integer, unless otherwise specified.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures, and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses, and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
- Unscheduled or unplanned readings will be presented within the participant's listings.
- Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be
  included in listings but omitted from figures (mean figures only for PK concentrations), summaries,
  and statistical analyses (excluding statistical analyses of PK parameters).

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables except for determining the worst-case values.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| | • |
|---|---|
| Descriptive Summary | y Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| <b>Graphical Displays</b> | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

### 10.3.3. Reporting Standards for Pharmacokinetics

| • | |
|---|---|
| Pharmacokinetic Con | centration Data |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. For continuous data: NQs at the beginning of a participant profile (i.e. before the first incidence of a measurable concentration) are deemed to be zero as it is assumed that in this circumstance no drug is yet measurable in the blood. For NQs at the end of the participant profile (i.e. after the last incidence of a measurable concentration); for individual plots and PK analyses these are dropped (set to missing) as they do not provide any useful information (and can erroneously indicate that absolutely no drug is present) for summary statistics, these are set to 0 (to avoid skewing of the summary statistics) Individual NQs which fall between two measurable concentrations are set to missing (individual values of this nature are assumed to be an anomaly) If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual participant plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the derivation of pharmacokinetic parameters, these NQs and any subsequent measurable concentrations will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Para | ameter Data |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | N, n, arithmetic mean, 95% CI of arithmetic mean, geometric mean, 95% CI of geometric mean, SD, SD of log (ln) data, CV (%), and between-subject geometric coefficient of variation (CVb (%)) will be reported. $ \text{CV}_b \text{ (%)} = \sqrt{\left(\text{exp}(\text{SD}^2) - 1\right) * 100} $ (SD[ln] = SD of Ln-Transformed data) |


| Parameters Not<br>Being Ln-<br>Transformed | Tmax, λz, λz lower, λz upper, and λz no. of points. |
|---|---|
| Parameters Not<br>Being Summarized | λz, λz lower, λz upper, and λz no. of points. |
| Listings | Include the first point, last point and number of points used in the determination of $\lambda z$ and Rsq_adjusted for listings. |

### 10.4. Appendix 4: Derived and Transformed Data

#### 10.4.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- The worst finding/interpretation associated with multiple measurements as the finding/interpretation for that time point.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from Dose Date on Day 1:
  - Assessment Date = Missing
    - → Study Day = Missing
    - Assessment Date < Dose Date on Day 1
      - → Study Day = Assessment Date –Dose Date on Day 1
  - Assessment Date >= Dose Date on Day 1
    - → Study Day = Assessment Date Dose Date on Day 1 + 1

#### 10.4.2. Study Population

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing day will have this imputed as day '15'.
  - o Any participant with a missing day and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### 10.4.3. Safety

#### **Adverse Events**

#### **AEs of Special Interest**

- QT prolongation
- Gastrointestinal intolerability and gastric toxicity
- Psychiatric events
- Nervous system disorders
- Skin and subcutaneous tissue disorders

### 12-Lead Electrocardiograms

#### QTcB Interval

• QTcB interval in msec will be calculated using QT interval (msec) and RR interval (msec) as

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

where RR interval in msec is calculated using QT interval (msec) and QTcF interval (msec) as

$$RR = (\frac{QT}{QTcF})^3 \times 1000$$

# 10.5. Appendix 5: Reporting Standards for Missing Data

# 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e., as specified in the protocol) is defined as the participant has completed all phases of the study including the final date on which data were or are expected to be collected.</li> <li>Withdrawn participants will not be replaced in the study.</li> <li>All available data from participants who are withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

### 10.5.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Section 10.2.2.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the eCRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a "01" will be used for the day and "Jan" will be used for the month</li> <li>If the partial date is a stop date, a "28/29/30/31" will be used for the day (dependent on the month and year) and "Dec" will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.6. Appendix 6: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events

### 10.6.1. Laboratory Values

Laboratory abnormalities will be graded according to the DAIDS grading table Version 2.1, July 2017. Laboratory results are converted to use SI units; only the numeric part of the criteria will be used. If for a laboratory parameter there are multiple grades sharing the same criteria, the maximum grade will be used.



| CCI - Th | nis secti | on contained | Clinical | Outcome / | Assessme | ent data c | collection | ı questior | nnaires or | indices, | , which | are prote | ected by t | hird pa | rty copyrig | jht laws a | ind |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| therefor | e have | on contained<br>been exclude | ed. | | | | | | | | | | | | | | |


| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and |
|---|
| therefore have been excluded. |

# 10.7. Appendix 7: Values of Potential Clinical Importance

# 10.7.1. ECG

| ECG Parameter | Units | Potential Clinical | Potential Clinically Important Range |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | · |
| Absolute QTc Interval | msec | | >450 |
| Absolute PR Interval | msec | <110 | >200 |
| Absolute QRS Interval | msec | <b>&lt;7</b> 5 | >110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | >60 |

# 10.7.2. Vital Signs

| Vital Sign Parameter | Units | Potential Clinically Important Range | |
|---|---|---|---|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | <85 | >140 |
| Diastolic Blood Pressure | mmHg | <45 | >90 |
| Heart Rate | Beats per<br>minute | <40 | >100 |

# 10.8. Appendix 8: Abbreviations & Trademarks

# 10.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | analysis data model |
| AE | adverse event |
| ALT | alanine aminotransferase |
| AUC | area under the plasma concentration-time curve |
| AUC(0-τ) | AUC from time 0 to the end of the dosing interval at steady state |
| BID | twice daily |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | confidence interval |
| Cmax | maximum observed concentration |
| CSR | clinical study report |
| C-SSRS | Columbia suicide severity rating scale |
| Сτ | plasma concentration at the end of the dosing interval |
| CV <sub>b</sub> | coefficient of variation (between) |
| CVw | coefficient of variability (within) |
| DAIDS | division of AIDS |
| DBF | database freeze |
| DBR | database release |
| DP | decimal places |
| DRV | darunavir |
| ECG | electrocardiogram |
| eCRF | electronic case record form |
| GSK | GlaxoSmithKline |
| ETR | etravirine |
| HIV | human immunodeficiency virus |
| ICH | international conference on harmonization |
| IDSL | integrated data standards library |
| LLN | lower limit of normal |
| NQ | not quantifiable |
| PK | pharmacokinetic |
| QD | once daily |
| RAP | reporting & analysis plan |
| SAC | statistical analysis complete |
| SAE | serious adverse event |
| SD | standard deviation |
| SDTM | study data tabulation model |
| SMQ | Standardized MedDRA Query |
| Tmax | time of maximum observed concentration |
| ULN | upper limit of normal |

# 10.8.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of |
|--------------------------------------------|
| Companies |
| NONE |

| Trademarks not owned by the GlaxoSmithKline |
|---------------------------------------------|
| Group of Companies |

SAS

WinNonlin

### 10.9. Appendix 9: List of Data Displays

### 10.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.8 | |
| Safety | 2.1 to 2.30 | 2.1 to 2.1 |
| Pharmacokinetic | 3.1 to 3.42 | 3.1 to 3.45 |
| Section | Listi | ngs |
| ICH Listings | 1 to | 32 |
| Non-ICH Listings | 33 to | 43 |

### 10.9.2. Mock Example Shell Referencing

Non-IDSL specifications will be referenced as indicated and if required example mock-up displays provided in the Table/Listing/Figure Shells.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

 Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.9.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

# 10.9.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | Subject Disposition | | | | |
| 1.1. | Enrolled | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | | SAC |
| 1.2. | Screened | SP1 | Summary of Study Population | | SAC |
| 1.3. | Safety | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | | SAC |
| 1.4. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failures | | SAC |
| Protoc | ol Deviation | | | , | , |
| 1.5. | Safety | DV1 | Summary of Important Protocol Deviations | | SAC |
| Demog | Demographic and Baseline Characteristics | | | | |
| 1.6. | Safety | DM1 | Summary of Demographic Characteristics | | SAC |
| 1.7. | Safety | DM5 | Summary of Race and Racial Combinations | | SAC |
| 1.8. | Safety | DM11 | Summary of Age Ranges | | SAC |

# 10.9.5. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 2.1. | Safety | AE1CP | Summary of Adverse Events by System Organ Class and Preferred Term | | SAC |
| 2.2. | Safety | AE1CP | Summary of Drug-Related Adverse Events by System Organ Class and Preferred Term | | SAC |
| 2.3. | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency | | SAC |
| 2.4. | Safety | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| 2.5. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| 2.6. | Safety | AE5A | Summary of Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | | SAC |
| 2.7. | Safety | AE1CP | Summary of Adverse Events of Special Interest | | SAC |
| Labora | tory: Chemistry | 1 | | | |
| 2.8. | Safety | LB1 | Summary of Clinical Chemistry Changes from Baseline | | SAC |
| 2.9. | Safety | LB1 | Summary of Clinical Chemistry Values | | SAC |
| 2.10. | Safety | LB16 | Summary of Clinical Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline | | SAC |
| _abora | tory: Hematolo | gy | | | |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.11. | Safety | LB1 | Summary of Hematology Changes from Baseline | | SAC |
| 2.12. | Safety | LB1 | Summary of Hematology Values | | SAC |
| 2.13. | Safety | LB16 | Summary of Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline | | SAC |
| Labora | tory: Urinalysis | <b>3</b> | | | |
| 2.14. | Safety | UR3 | Summary of Urinalysis Dipstick Results | | SAC |
| 2.15. | Safety | LB1 | Summary of Urine Concentration Changes from Baseline | | SAC |
| 2.16. | Safety | LB1 | Summary of Urine Concentration Values | | SAC |
| 2.17. | Safety | LB16 | Summary of Urinalysis by Maximum Grade Increase Post-<br>Baseline Relative to Baseline | | SAC |
| ECG | | | | | |
| 2.18. | Safety | SAFE_T1 | Summary of ECG Findings | | SAC |
| 2.19. | Safety | EG2 | Summary of ECG Changes from Baseline | | SAC |
| 2.20. | Safety | EG2 | Summary of ECG Values | | SAC |
| 2.21. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| 2.22. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| Vital Si | gns | | | | • |
| 2.23. | Safety | VS1 | Summary of Vital Sign Changes from Baseline | | SAC |
| 2.24. | Safety | VS1 | Summary of Vital Sign Values | | SAC |
| C-SSRS | 3 | | | 1 | 1 |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.25. | Safety | CSSRS4 | Listing of C-SSRS Suicidal Ideation and Behaviour Data | Only include participants who have suicidal ideation or behaviour | SAC |
| Liver E | vent | | | | |
| 2.26. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | | SAC |
| 2.27. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | | SAC |
| COVID- | 19 Related AE | | | | |
| 2.28. | Safety | PAN1 | Summary of COVID-19 Assessment | | SAC |
| 2.29 | Safety | SAFE_T2 | Summary of COVID-19 Adverse Event | | SAC |
| 2.30 | Safety | PAN11 | Summary of COVID-19 Symptoms for Subjects with Adverse Events | Conditional Display | SAC |

# 10.9.6. Safety Figures

| Safety: F | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | | | | | |
| 2.1. | Safety | EG9 | Mean (95% CI) Change from Baseline in QTcF Interval by Timepoint and Treatment | | SAC |

### 10.9.7. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| PK Cor | centration Data | | | | |
| 3.1. | PK<br>Concentration | PKCT1 | Summary of GSK3640254 Plasma Pharmacokinetic Concentration-Time Data (units) by Treatment – Cohort 1 | | SAC |
| 3.2. | PK<br>Concentration | PKCT1 | Summary of Darunavir Plasma Pharmacokinetic Concentration-<br>Time Data (units) by Treatment – Cohort 1 | | SAC |
| 3.3. | PK<br>Concentration | PKCT1 | Summary of Ritonavir Plasma Pharmacokinetic Concentration-<br>Time Data (units) by Treatment – Cohort 1 | | SAC |
| 3.4. | PK<br>Concentration | PKCT1 | Summary of Predose (trough) GSK3640254 Plasma<br>Concentration Data (units) by Treatment – Cohort 1 | | SAC |
| 3.5. | PK<br>Concentration | PKCT1 | Summary of Predose (trough) Darunavir Plasma Concentration Data (units) by Treatment – Cohort 1 | | SAC |
| 3.6. | PK<br>Concentration | PKCT1 | Summary of Predose (trough) Ritonavir Plasma Concentration Data (units) by Treatment – Cohort 1 | | SAC |
| 3.7. | PK<br>Concentration | PKCT1 | Summary of GSK3640254 Plasma Pharmacokinetic Concentration-Time Data (units) by Treatment – Cohort 2 | | SAC |
| 3.8. | PK<br>Concentration | PKCT1 | Summary of Etravirine Plasma Pharmacokinetic Concentration-<br>Time Data (units) by Treatment – Cohort 2 | | SAC |
| 3.9. | PK<br>Concentration | PKCT1 | Summary of Predose (trough) GSK3640254 Plasma<br>Concentration Data (units) by Treatment – Cohort 2 | | SAC |
| 3.10. | PK<br>Concentration | PKCT1 | Summary of Predose (trough) Etravirine Plasma Concentration Data (units) by Treatment – Cohort 2 | | SAC |
| 3.11. | PK<br>Concentration | PKCT1 | Summary of GSK3640254 Plasma Pharmacokinetic Concentration-Time Data (units) by Treatment – Cohort 3 | | SAC |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.12. | PK<br>Concentration | PKCT1 | Summary of Darunavir Plasma Pharmacokinetic Concentration-<br>Time Data (units) by Treatment – Cohort 3 | | SAC |
| 3.13. | PK<br>Concentration | PKCT1 | Summary of Ritonavir Plasma Pharmacokinetic Concentration-<br>Time Data (units) by Treatment – Cohort 3 | | SAC |
| 3.14. | PK<br>Concentration | PKCT1 | Summary of Etravirine Plasma Pharmacokinetic Concentration-<br>Time Data (units) by Treatment – Cohort 3 | | SAC |
| 3.15. | PK<br>Concentration | PKCT1 | Summary of Predose (trough) GSK3640254 Plasma<br>Concentration Data (units) by Treatment – Cohort 3 | | SAC |
| 3.16. | PK<br>Concentration | PKCT1 | Summary of Predose (trough) Darunavir Plasma Concentration Data (units) by Treatment – Cohort 3 | | SAC |
| 3.17. | PK<br>Concentration | PKCT1 | Summary of Predose (trough) Ritonavir Plasma Concentration Data (units) by Treatment – Cohort 3 | | SAC |
| 3.18. | PK<br>Concentration | PKCT1 | Summary of Predose (trough) Etravirine Plasma Concentration Data (units) by Treatment – Cohort 3 | | SAC |
| PK Der | ived Parameters | ; | | | |
| 3.19. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived GSK3640254 Plasma Pharmacokinetic Parameters (Non-Transformed) Based on Actual Time by Treatment – Cohort 1 | | SAC |
| 3.20. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived GSK3640254 Plasma Pharmacokinetic Parameters (Ln-Transformed) Based on Actual Time by Treatment – Cohort 1 | | SAC |
| 3.21. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Darunavir Plasma Pharmacokinetic Parameters (Non-Transformed) Based on Actual Time by Treatment – Cohort 1 | | SAC |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.22. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Darunavir Plasma Pharmacokinetic Parameters (Ln-Transformed) Based on Actual Time by Treatment – Cohort 1 | | SAC |
| 3.23. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Ritonavir Plasma Pharmacokinetic Parameters (Non-Transformed) Based on Actual Time by Treatment – Cohort 1 | | SAC |
| 3.24. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Ritonavir Plasma Pharmacokinetic Parameters (Ln-Transformed) Based on Actual Time by Treatment – Cohort 1 | | SAC |
| 3.25. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived GSK3640254 Plasma Pharmacokinetic Parameters (Non-Transformed) Based on Actual Time by Treatment – Cohort 2 | | SAC |
| 3.26. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived GSK3640254 Plasma Pharmacokinetic Parameters (Ln-Transformed) Based on Actual Time by Treatment – Cohort 2 | | SAC |
| 3.27. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Etravirine Plasma Pharmacokinetic Parameters (Non-Transformed) Based on Actual Time by Treatment – Cohort 2 | | SAC |
| 3.28. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Etravirine Plasma Pharmacokinetic Parameters (Ln-Transformed) Based on Actual Time by Treatment – Cohort 2 | | SAC |
| 3.29. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived GSK3640254 Plasma Pharmacokinetic Parameters (Non-Transformed) Based on Actual Time by Treatment – Cohort 3 | | SAC |
| 3.30. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived GSK3640254 Plasma Pharmacokinetic Parameters (Ln-Transformed) Based on Actual Time by Treatment – Cohort 3 | | SAC |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.31. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Darunavir Plasma Pharmacokinetic Parameters (Non-Transformed) Based on Actual Time by Treatment – Cohort 3 | | SAC |
| 3.32. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Darunavir Plasma Pharmacokinetic Parameters (Ln-Transformed) Based on Actual Time by Treatment – Cohort 3 | | SAC |
| 3.33. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Ritonavir Plasma Pharmacokinetic Parameters (Non-Transformed) Based on Actual Time by Treatment – Cohort 3 | | SAC |
| 3.34. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Ritonavir Plasma Pharmacokinetic Parameters (Ln-Transformed) Based on Actual Time by Treatment – Cohort 3 | | SAC |
| 3.35. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Etravirine Plasma Pharmacokinetic Parameters (Non-Transformed) Based on Actual Time by Treatment – Cohort 3 | | SAC |
| 3.36. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Etravirine Plasma Pharmacokinetic Parameters (Ln-Transformed) Based on Actual Time by Treatment – Cohort 3 | | SAC |
| PK Ana | lysis Tables | | | | |
| 3.37. | PK<br>Parameter | PKPT3 | Statistical Analysis of GSK3640254 Plasma Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Cohort 1 | AUC(0-tau) and Cmax | SAC |
| 3.38. | PK<br>Parameter | PKPT3 | Statistical Analysis of Darunavir Plasma Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Cohort 1 | AUC(0-tau) and Cmax | SAC |
| 3.39. | PK<br>Parameter | PKPT3 | Statistical Analysis of Ritonavir Plasma Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Cohort 1 | AUC(0-tau) and Cmax | SAC |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.40. | PK<br>Parameter | PKPT3 | Statistical Analysis of GSK3640254 Plasma Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Cohort 2 | AUC(0-tau) and Cmax | SAC |
| 3.41. | PK<br>Parameter | PKPT3 | Statistical Analysis of Etravirine Plasma Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Cohort 2 | AUC(0-tau) and Cmax | SAC |
| 3.42. | PK<br>Parameter | PKPT3 | Statistical Analysis of GSK3640254 Plasma Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Cohort 3 | AUC(0-tau) and Cmax | SAC |

# 10.9.8. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individ | ual Concentration | on Plots | | | • |
| 3.1. | PK<br>Concentration | PKCF1 | Individual GSK3640254 Plasma Concentration-Time Plots by Participant – Cohort 1 (Linear and Semi-Logarithmic) | Paginate by Participant Dashed line represents the LLQ Treatments Overlaid | SAC |
| 3.2. | PK<br>Concentration | PKCF1 | Individual Darunavir Plasma Concentration-Time Plots by Participant – Cohort 1 (Linear and Semi-Logarithmic) | Paginate by Participant Dashed line represents the LLQ Treatments Overlaid | SAC |
| 3.3. | PK<br>Concentration | PKCF1 | Individual Ritonavir Plasma Concentration-Time Plots by Participant – Cohort 1 (Linear and Semi-Logarithmic) | Paginate by Participant Dashed line represents the LLQ Treatments Overlaid | SAC |
| 3.4. | PK<br>Concentration | PKCF1 | Individual GSK3640254 Plasma Concentration-Time Plots by Treatment – Cohort 1 (Linear and Semi-Logarithmic) | Paginate by Treatment Dashed line represents the LLQ Participants Overlaid | SAC |
| 3.5. | PK<br>Concentration | PKCF1 | Individual Darunavir Plasma Concentration-Time Plots by Treatment – Cohort 1 (Linear and Semi-Logarithmic) | Paginate by Treatment Dashed line represents the LLQ Participants Overlaid | SAC |
| 3.6. | PK<br>Concentration | PKCF1 | Individual Ritonavir Plasma Concentration-Time Plots by Treatment – Cohort 1 (Linear and Semi-Logarithmic) | Paginate by Treatment Dashed line represents the LLQ Participants Overlaid | SAC |
| 3.7. | PK<br>Concentration | PKCF1 | Individual GSK3640254 Plasma Concentration-Time Plots by Participant – Cohort 2 (Linear and Semi-Logarithmic) | Paginate by Participant Dashed line represents the LLQ Treatments Overlaid | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.8. | PK<br>Concentration | PKCF1 | Individual Etravirine Plasma Concentration-Time Plots by Participant – Cohort 2 (Linear and Semi-Logarithmic) | Paginate by Participant Dashed line represents the LLQ Treatments Overlaid | SAC |
| 3.9. | PK<br>Concentration | PKCF1 | Individual GSK3640254 Plasma Concentration-Time Plots by Treatment – Cohort 2 (Linear and Semi-Logarithmic) | Paginate by Treatment Dashed line represents the LLQ Participants Overlaid | SAC |
| 3.10. | PK<br>Concentration | PKCF1 | Individual Etravirine Plasma Concentration-Time Plots by Treatment – Cohort 2 (Linear and Semi-Logarithmic) | Paginate by Treatment Dashed line represents the LLQ Participants Overlaid | SAC |
| 3.11. | PK<br>Concentration | PKCF1 | Individual GSK3640254 Plasma Concentration-Time Plots by Participant – Cohort 3 (Linear and Semi-Logarithmic) | Paginate by Participant Dashed line represents the LLQ Treatments Overlaid | SAC |
| 3.12. | PK<br>Concentration | PKCF1 | Individual Darunavir Plasma Concentration-Time Plots by Participant – Cohort 3 (Linear and Semi-Logarithmic) | Paginate by Participant Dashed line represents the LLQ | SAC |
| 3.13. | PK<br>Concentration | PKCF1 | Individual Ritonavir Plasma Concentration-Time Plots by Participant – Cohort 3 (Linear and Semi-Logarithmic) | Paginate by Participant Dashed line represents the LLQ | SAC |
| 3.14. | PK<br>Concentration | PKCF1 | Individual Etravirine Plasma Concentration-Time Plots by Participant – Cohort 3 (Linear and Semi-Logarithmic) | Paginate by Participant Dashed line represents the LLQ | SAC |
| 3.15. | PK<br>Concentration | PKCF1 | Individual GSK3640254 Plasma Concentration-Time Plots by Treatment – Cohort 3 (Linear and Semi-Logarithmic) | Paginate by Treatment Dashed line represents the LLQ Participants Overlaid | SAC |
| 3.16. | PK<br>Concentration | PKCF1 | Individual Darunavir Plasma Concentration-Time Plots by Treatment – Cohort 3 (Linear and Semi-Logarithmic) | Dashed line represents the LLQ Participants Overlaid | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.17. | PK<br>Concentration | PKCF1 | Individual Ritonavir Plasma Concentration-Time Plots by Treatment – Cohort 3 (Linear and Semi-Logarithmic) | Dashed line represents the LLQ Participants Overlaid | SAC |
| 3.18. | PK<br>Concentration | PKCF1 | Individual Etravirine Plasma Concentration-Time Plots by Treatment – Cohort 3 (Linear and Semi-Logarithmic) | Dashed line represents the LLQ Participants Overlaid | SAC |
| Mean / | Median Concen | tration Plots | | | • |
| 3.19. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) GSK3640254 Plasma Concentration-Time Plots by Treatment – Cohort 1 (Linear and Semi-Logarithmic) | Treatments Overlaid | SAC |
| 3.20. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Darunavir Plasma Concentration-<br>Time Plots by Treatment – Cohort 1 (Linear and Semi-<br>Logarithmic) | Treatments Overlaid | SAC |
| 3.21. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Ritonavir Plasma Concentration-<br>Time Plots by Treatment – Cohort 1 (Linear and Semi-<br>Logarithmic) | Treatments Overlaid | SAC |
| 3.22. | PK<br>Concentration | PKCF3 | Median (Range) GSK3640254 Plasma Concentration-Time Plots by Treatment – Cohort 1 (Linear and Semi-Logarithmic) | Treatments Overlaid | SAC |
| 3.23. | PK<br>Concentration | PKCF3 | Median (Range) Darunavir Plasma Concentration-Time Plots by Treatment – Cohort 1 (Linear and Semi-Logarithmic) | Treatments Overlaid | SAC |
| 3.24. | PK<br>Concentration | PKCF3 | Median (Range) Ritonavir Plasma Concentration-Time Plots by Treatment – Cohort 1 (Linear and Semi-Logarithmic) | Treatments Overlaid | SAC |
| 3.25. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Predose (Trough) GSK3640254 Plasma Concentration-Time Plots by Treatment – Cohort 1 (Linear and Semi-Logarithmic) | | SAC |
| 3.26. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Predose (Trough) Darunavir Plasma<br>Concentration-Time Plots by Treatment – Cohort 1 (Linear and<br>Semi-Logarithmic) | | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.27. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Predose (Trough) Ritonavir Plasma<br>Concentration-Time Plots by Treatment – Cohort 1 (Linear and<br>Semi-Logarithmic) | | SAC |
| 3.28. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) GSK3640254 Plasma Concentration-Time Plots by Treatment – Cohort 2 (Linear and Semi-Logarithmic) | Treatments Overlaid | SAC |
| 3.29. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Etravirine Plasma Concentration-<br>Time Plots by Treatment – Cohort 2 (Linear and Semi-<br>Logarithmic) | Treatments Overlaid | SAC |
| 3.30. | PK<br>Concentration | PKCF3 | Median (Range) GSK3640254 Plasma Concentration-Time Plots by Treatment – Cohort 2 (Linear and Semi-Logarithmic) | Treatments Overlaid | SAC |
| 3.31. | PK<br>Concentration | PKCF3 | Median (Range) Etravirine Plasma Concentration-Time Plots by Treatment – Cohort 2 (Linear and Semi-Logarithmic) | Treatments Overlaid | SAC |
| 3.32. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Predose (Trough) GSK3640254 Plasma Concentration-Time Plots by Treatment – Cohort 2 (Linear and Semi-Logarithmic) | | SAC |
| 3.33. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Predose (Trough) Etravirine Plasma Concentration-Time Plots by Treatment – Cohort 2 (Linear and Semi-Logarithmic) | | SAC |
| 3.34. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) GSK3640254 Plasma Concentration-Time Plots by Treatment – Cohort 3 (Linear and Semi-Logarithmic) | Treatments Overlaid | SAC |
| 3.35. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Darunavir Plasma Concentration-<br>Time Plots by Treatment – Cohort 3 (Linear and Semi-<br>Logarithmic) | | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.36. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Ritonavir Plasma Concentration-<br>Time Plots by Treatment – Cohort 3 (Linear and Semi-<br>Logarithmic) | | SAC |
| 3.37. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Etravirine Plasma Concentration-<br>Time Plots by Treatment – Cohort 3 (Linear and Semi-<br>Logarithmic) | | SAC |
| 3.38. | PK<br>Concentration | PKCF3 | Median (Range) GSK3640254 Plasma Concentration-Time Plots by Treatment – Cohort 3 (Linear and Semi-Logarithmic) | Treatments Overlaid | SAC |
| 3.39. | PK<br>Concentration | PKCF3 | Median (Range) Darunavir Plasma Concentration-Time Plots by Treatment – Cohort 3 (Linear and Semi-Logarithmic) | | SAC |
| 3.40. | PK<br>Concentration | PKCF3 | Median (Range) Ritonavir Plasma Concentration-Time Plots by Treatment – Cohort 3 (Linear and Semi-Logarithmic) | | SAC |
| 3.41. | PK<br>Concentration | PKCF3 | Median (Range) Etravirine Plasma Concentration-Time Plots by Treatment – Cohort 3 (Linear and Semi-Logarithmic) | | SAC |
| 3.42. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Predose (Trough) GSK3640254 Plasma Concentration-Time Plots by Treatment – Cohort 3 (Linear and Semi-Logarithmic) | | SAC |
| 3.43. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Predose (Trough) Darunavir Plasma<br>Concentration-Time Plots by Treatment – Cohort 3 (Linear and<br>Semi-Logarithmic) | | SAC |
| 3.44. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Predose (Trough) Ritonavir Plasma<br>Concentration-Time Plots by Treatment – Cohort 3 (Linear and<br>Semi-Logarithmic) | | SAC |
| 3.45. | PK<br>Concentration | PKCF2 | Mean (Standard Deviation) Predose (Trough) Etravirine Plasma<br>Concentration-Time Plots by Treatment – Cohort 3 (Linear and<br>Semi-Logarithmic) | | SAC |

# 10.9.9. ICH Listings

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | , |
| 1. | Safety | ES3 | Listing of Reasons for Study Withdrawal | | SAC |
| 2. | Safety | SD2 | Listing of Reasons for Study Treatment Discontinuation | | SAC |
| 3. | Screened | ES7 | Listing of Reasons for Screen Failure | | SAC |
| Protoco | l Deviations | | | | • |
| 4. | Safety | DV2 | Listing of Important Protocol Deviations | | SAC |
| 5. | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Populat | ions Analyzed | | | | |
| 6. | Safety | SP3A | Listing of Subjects Excluded from Any Population | | SAC |
| Demog | raphic and Bas | seline Characteris | tics | | • |
| 7. | Safety | DM2 | Listing of Demographic Characteristics | | SAC |
| 8. | Safety | DM9 | Listing of Race | | SAC |
| Prior ar | nd Concomitan | t Medications | | | • |
| 9. | Safety | CM5 | Listing of Concomitant Medications | Based on GSK Drug Dictionary | SAC |
| Exposu | re and Treatme | ent Compliance | | | |
| 10. | Safety | EX4 | Listing of Exposure Data | | SAC |
| 11. | Safety | POP_L1 | Listing of Meal Data | | SAC |
| Adverse | e Events | | | | |
| 12. | Safety | AE2 | Listing of Relationship Between System Organ Class and Verbatim Text | | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 13. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 14. | Safety | AE9CP | Listing of All Adverse Events | | SAC |
| 15. | Safety | AE9CP | Listing of Adverse Events of Special Interest | | SAC |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 16. | Safety | AE9CP | Listing of Study Drug Related Adverse Events | | SAC |
| 17. | Safety | AE9CP | Listing of Serious Adverse Events (Fatal & Non-Fatal) | | SAC |
| 18. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | SAC |
| 19. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study | | SAC |
| Hepato | biliary (Liver) | | | | |
| 20. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events | | SAC |
| 21. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | | SAC |
| All Lab | oratory | | | | |
| 22. | Safety | LB5A | Listing of Clinical Chemistry with any Toxicities | | SAC |
| 23. | Safety | LB5A | Listing of All Clinical Chemistry Data for Subjects with any Toxicities | | SAC |
| 24. | Safety | LB5A | Listing of Hematology with any Toxicities | | SAC |
| 25. | Safety | LB5A | Listing of All Hematology Data for Subjects with any Toxicities | | SAC |
| 26. | Safety | LB5A | Listing of Urinalysis with any Toxicities | | SAC |
| 27. | Safety | LB5A | Listing of All Urinalysis Data for Subjects with any Toxicities | | SAC |
| ECG | | | | | |
| 28. | Safety | EG6 | Listing of All ECG Findings | | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 29. | Safety | EG6 | Listing of All Abnormal ECG Findings | | SAC |
| 30. | Safety | EG4 | Listing of All ECG Values | | SAC |
| Vital Sig | gns | | | | |
| 31. | Safety | VS5 | Listing of All Vital Signs of Potential Clinical Importance | | SAC |
| 32. | Safety | VS5 | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance | | SAC |

# 10.9.10. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Pharm | acokinetics | | | | |
| 33. | PK<br>Concentration | PKCL1P | Listing of GSK3640254 Plasma Concentrations (ng/mL) by Treatment – Cohort 1 | | SAC |
| 34. | PK<br>Concentration | PKCL1P | Listing of Darunavir Plasma Concentrations (ng/mL) by Treatment – Cohort 1 | | SAC |
| 35. | PK<br>Concentration | PKCL1P | Listing of Ritonavir Plasma Concentrations (ng/mL) by Treatment – Cohort 1 | | SAC |
| 36. | PK Parameter | PKPL1P | Listing of GSK3640254 Plasma Pharmacokinetic Parameters Based on Actual Time by Treatment – Cohort 1 | | SAC |
| 37. | PK Parameter | PKPL1P | Listing of Darunavir Plasma Pharmacokinetic Parameters Based on Actual Time by Treatment – Cohort 1 | | SAC |
| 38. | PK Parameter | PKPL1P | Listing of Ritonavir Plasma Pharmacokinetic Parameters Based on Actual Time by Treatment – Cohort 1 | | SAC |
| 39. | PK<br>Concentration | PKCL1P | Listing of GSK3640254 Plasma Concentrations (ng/mL) by Treatment – Cohort 2 | | SAC |
| 40. | PK<br>Concentration | PKCL1P | Listing of Etravirine Plasma Concentrations (ng/mL) by Treatment – Cohort 2 | | SAC |
| 41. | PK Parameter | PKPL1P | Listing of GSK3640254 Plasma Pharmacokinetic Parameters Based on Actual Time by Treatment – Cohort 2 | | SAC |
| 42. | PK Parameter | PKPL1P | Listing of Etravirine Plasma Pharmacokinetic Parameters Based on Actual Time by Treatment – Cohort 2 | | SAC |
| 43. | PK<br>Concentration | PKCL1P | Listing of GSK3640254 Plasma Concentrations (ng/mL) by Treatment – Cohort 3 | | SAC |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 44. | PK<br>Concentration | PKCL1P | Listing of Darunavir Plasma Concentrations (ng/mL) by Treatment – Cohort 3 | | SAC |
| 45. | PK<br>Concentration | PKCL1P | Listing of Ritonavir Plasma Concentrations (ng/mL) by Treatment – Cohort 3 | | SAC |
| 46. | PK<br>Concentration | PKCL1P | Listing of Etravirine Plasma Concentrations (ng/mL) by Treatment – Cohort 3 | | SAC |
| 47. | PK Parameter | PKPL1P | Listing of GSK3640254 Plasma Pharmacokinetic Parameters Based on Actual Time by Treatment – Cohort 3 | | SAC |
| 48. | PK Parameter | PKPL1P | Listing of Darunavir Plasma Pharmacokinetic Parameters Based on Actual Time by Treatment – Cohort 3 | | SAC |
| 49. | PK Parameter | PKPL1P | Listing of Ritonavir Plasma Pharmacokinetic Parameters Based on Actual Time by Treatment – Cohort 3 | | SAC |
| 50. | PK Parameter | PKPL1P | Listing of Etravirine Plasma Pharmacokinetic Parameters Based on Actual Time by Treatment – Cohort 3 | | SAC |
| 51. | Safety | PAN12 | Listing of COVID-19 Assessments and Symptom Assessment | | SAC |
| 52. | Safety | AE9CP | Listing of Adverse Events of COVID-19 | | SAC |